CLINICAL TRIAL: NCT01392586
Title: Systemic Therapy With or Without Up Front Surgery of the Primary Tumor in Breast Cancer Patients With Distant Metastases at Initial presenTation
Brief Title: Systemic Therapy With or Without Upfront Surgery in Metastatic Breast Cancer
Acronym: SUBMIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to low accrual rate
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Principal Investigator, M.F. Ernst, dr, Dr.M.F.Ernst, Jeroen Bosch Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2010-05
Record Dates: First submitted 2011-07-05; First posted 2011-07-12 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Breast Cancer
Keywords: survival; systemic therapy; upfront surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upfront surgery (Experimental): Upfront surgery followed by systemic treatment
  Interventions: Procedure: upfront breast surgery
- Systemic therapy (Other): Systemic therapy possibly followed by local treatment of the breast tumor
  Interventions: Other: systemic therapy

INTERVENTIONS:
Procedure: upfront breast surgery — surgery of primary tumor, lumpectomy or mastectomy
  Arms: Upfront surgery
Other: systemic therapy — chemotherapy, immunotherapy or endocrine therapy (possibly followed by local surgery of the breast)
  Arms: Systemic therapy

SUMMARY:
SUBMIT is a clinical trial that intends to answer the question whether up front breast surgery in patients with primary distant metastatic breast cancer will result in an improvement of the 2-year survival compared to the survival achieved with systemic therapy and delayed local treatment or systemic therapy alone.

Randomization will take place immediately after the diagnosis of primary distant metastatic breast cancer. Patients either randomize for up front surgery of the breast tumor (UFS) followed by systemic therapy or for systemic therapy (ST) potentially followed by delayed local treatment of the breast tumor.

The primary endpoint of this trial is the 2-years survival. Quality of life is one of the most important secondary endpoints.

DETAILED DESCRIPTION:
In the Netherlands approximately one out of eight women will be diagnosed with breast cancer; 5% have metastatic disease at presentation. Because metastatic breast cancer is considered to be an incurable disease, it is only treated with a palliative intent. Recent retrospective studies have demonstrated that (complete) resection of the primary tumor significantly improves the outcome of patients with primary metastatic breast cancer. However, other studies showed that the survival benefit in patients who underwent surgery is caused by selection bias.

SUBMIT is a clinical trial that intends to answer the question whether up front breast surgery in patients with primary distant metastatic breast cancer will result in an improvement of the 2-year survival compared to the survival achieved with systemic therapy and delayed local treatment or systemic therapy alone.

Patients to submit in this study are patients with primary distant metastatic breast cancer, with no prior treatment of the breast cancer, who are 18 years or older and fit enough to undergo surgery and systemic therapy. Exclusion criteria are: history of breast cancer, other malignancy within the last 10 years, surgical treatment or radiotherapy of this breast tumor before randomization, irresectable T4 tumor or synchronous bilateral breastcancer.

Randomization will take place immediately after the diagnosis of primary distant metastatic breast cancer. Patients either randomize for up front surgery of the breast tumor (UFS) followed by systemic therapy or for systemic therapy (ST) potentially followed by delayed local treatment of the breast tumor.

The primary endpoint of this trial is the 2-years survival. Quality of life is one of the most important secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed primary distant metastatic breast cancer (M1)
* Anticipated survival of at least 6 months
* Histologically proven breast cancer
* Hormonal and HER2Neu status should be known
* T1-T3, resectable T4 status, N0-N3
* Performance status of the patient should allow surgery / systemic therapy
* Co-morbidity of the patient should allow surgery / systemic therapy
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Primary invasive breast cancer in medical history
* Other malignancy within the last 10 years, besides basal cell carcinoma of the skin or early stage cervical cancer
* Surgical treatment / radiotherapy of this breast tumor before randomization
* Irresectable T4 breast tumor
* Synchronous bilateral breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Survival | participants will be followed until death (expected median survival 31 months for surgery group)
  Survival is defined in months from the time of randomization until death. Overall survival will be expressed as the median survival in months.

SECONDARY OUTCOMES:
Quality of Life | 5 years after randomisation
  The EORTC QLQ - C30 and BR23 questionnaires will be used for the measurement of the quality of life. The quality of life will be assessed at 3, 6, 12, 18 months and 2,3,4,5 years after randomisation
Two year survival | 2 yrs after randomisation
  The percentage of patients who survive two years after randomization will be determined.
Number of unplanned local therapies | 5-6 months after randomisation
  The number of patients who will receive local treatment at another point than scheduled
Difference in systemic therapy given | 6 months after randomisation
  register which patients receive what treatments
Determination of pathological resection margin | Pathological report approximately 1 day after surgery
  The definition of a complete resection in this trial means free resection margins for the invasive component.
Number of treatments of the axillary lymph nodes | 6 months after randomisation
  register which patients receive these treatments

CONTACTS AND LOCATIONS:
Overall Officials: M.F. Ernst, dr, Principal Investigator — Jeroen Bosch Ziekenhuis; A.C. Voogd, dr, Principal Investigator — Maastricht University Medical Centre; V.C.G. Tjan-Heijnen, Prof, dr, Principal Investigator — Maastricht University Medical Centre
Locations (26):
- Netherlands (26):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Wilhelmina Ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooiziekenhuizen, loc Blaricum, Blaricum
  - Reinier de Graaf, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Atrium Medisch Centrum, Heerlen
  - Ziekenhuis Elkerliek, loc Helmond, Helmond
  - Ziekenhuisgroep Twente, Loc. SMT, Hengelo
  - Spaarne Ziekenhuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Diaconessenhuis, Leiden
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Ziekenhuis, Loc. Nieuwegein, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - UMC St. Radboud, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Orbis Medisch Centrum, Sittard
  - Haga Ziekenhuis, Loc. Leijweg, The Hague
  - Ziekenhuis Bronovo, The Hague
  - St. Elisabeth Ziekenhuis, Tilburg
  - Viecuri Medisch Centrum, loc. St Maartens Gasthuis, Venlo
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Ruiterkamp J, Voogd AC, Tjan-Heijnen VC, Bosscha K, van der Linden YM, Rutgers EJ, Boven E, van der Sangen MJ, Ernst MF; Dutch Breast Cancer Trialists' Group (BOOG). SUBMIT: Systemic therapy with or without up front surgery of the primary tumor in breast cancer patients with distant metastases at initial presentation. BMC Surg. 2012 Apr 2;12:5. doi: 10.1186/1471-2482-12-5. PMID 22469291